







# **WATCH**Wessex AsThma CoHort of Difficult Asthma

## **VOLUNTEER CONSENT FORM**

| Do | cument Version: | 4.5,16 Feb 2018 | Study number: W_ | /_ |
|---|---|---|---|---|
| Eth | ics Rec No.: | 14/WM/1226 | | |
| Pri | ncipal Investigators: | Dr Ramesh Kurukulaaratchy, Pro | ofessor Peter Howartl | n |
| Bio<br>sha | This form is in three parts. Part A relates to the main WATCH study. Part B relates to the Detailed Biological Characterisation Sub-study. Part C is about storage of samples for genetic studies and data sharing. Please read all parts. You may consent to Part A, the main study, but not to Part B or C if you wish. | | | |
| Please initial one of the boxes against each statement, indicating whether you agree/consent or not. | | | | |
| PART A Consent for the main study. Agree / Consent? Yes No | | | | |
| 1. | this consent form; version WATCH and my part in it h | formation Sheet version 4.5, date 4.5, dated 16/02/2018. All make been answered and I have been to take part in this reseat | y questions about nad enough time to | |
| 2. | | rt is voluntary and that I am free son, and my medical care and or | | |
| 3. | my clinic visits, plus releva<br>other comparable GP heal<br>from University of Southam | sections of my medical notes, daint GP care data from Hampshire th record systems will be looked opton and from the UHS NHS Trustudy. I give permission for the control of | e Health Record or<br>I at by researchers<br>ust and included in | |
| 4. | from the inside of my mout collected, that giving samp | e samples to be taken and for sa<br>th and nose. I understand how t<br>les for this research is voluntary<br>to use of the samples at any tim<br>t be affected. | the samples will be and that I am free | |
| 5. | that they may ask for spu | nn, believes it will be helpful to my<br>tum (phlegm) samples. I agree<br>e samples may be stored and use | that, after this any | |
| 6. | that they may ask for a br | in, believes it will be helpful to my ronchoscopy. I agree that, after may be stored and used for research | this any remaining | |

| | | Agree / Consent? | | | |
|---|---|---|---|---|---|
| | | | | Yes | No |
| 7. | I understand that samples researchers at other academ are able to carry out analyse agree that samples collecte researchers. | ic institutions (hospita<br>s that will help resear | Is and universities) if they ch studies into asthma. I | | |
| 8. | I understand that samples<br>commercial companies (phare<br>out analyses that will help res<br>collected during this study may | maceutical companies<br>earch studies into astl | ) if they are able to carry nma. I agree that samples | | |
| 9. | I understand and agree that may be shared anonymously approved asthma research in may be in countries within or of that some of these countries transfer of personal data. I give | with other researchers<br>the future. I understa<br>outside the European l<br>outside the EEA do no | s to support other ethically<br>and that these researchers<br>Economic Area (EEA), and<br>of have laws regulating the | | |
| 10. I agree to my GP being informed of my participation in the study. I have informed you about my participation in any other research study. | | | | | |
| 11. | 11. I understand I shall not benefit financially if this research leads to the<br>development of a new treatment or test. | | | | |
| 12. | I understand I may be contact other local research studies. | cted in future to discus | ss possible participation in | | |
| Na | me of Patient | Date | Signature | · | |
| Nai | me of person taking consent | Date | -<br>Signature | | |

Page 2 of 5 WATCH study ICF Version 4.5, 16 Feb 2018. Ethics no. 14/WM/1226

One copy for patient, one for researcher, one to be kept with hospital notes.

## PART B Consent for Additional Biological Samples Agree / Consent? Yes 13. I have read the "Detailed Biological Characterisation" Patient Information Sheet version 1.0, dated 16/02/2018 and this consent form; version 4.5, dated 16/02/2018. All my questions about this WATCH sub study and my part in it have been answered and I have had enough time to make my decision. I freely consent to take part in this research study. 14. I agree for Exhaled Breath samples to be taken. I understand how the samples will be collected, that giving samples for this research is voluntary and that I am free to withdraw my agreement to use of the samples at any time, and my medical care and legal rights will not be affected. 15. I agree for Induced Sputum samples to be taken. I understand how the samples will be collected, that giving samples for this research is voluntary and that I am free to withdraw my agreement to use of the samples at any time, and my medical care and legal rights will not be affected. 16. I agree for Nasal Lavage samples to be taken. I understand how the samples will be collected, that giving samples for this research is voluntary and that I am free to withdraw my agreement to use of the samples at any time, and my medical care and legal rights will not be affected. 17. I agree for Nasal Brushing samples to be taken. I understand how the samples will be collected, that giving samples for this research is voluntary and that I am free to withdraw my agreement to use of the samples at any time, and my medical care and legal rights will not be affected. 18. I agree for Bronchoscopy samples to be taken. I understand how the samples will be collected, that giving samples for this research is voluntary and that I am free to withdraw my agreement to use of the samples at any time, and my medical care and legal rights will not be affected. I understand that undertaking this procedure will require a separate consent form, as required by UHS NHS Trust, at the time of the procedure. Name of Patient Date Signature

One copy for patient, one for researcher, one to be kept with hospital notes.

Date

Name of person taking consent

Signature

#### WATCH Volunteer Consent Form

### Part C Consent for storage of samples and participation in genetic studies/ genomic data sharing

We would also like to undertake some genetic analyses on the samples you have provided and to store any samples collected for future research in asthma. Genomic studies examine genetic differences across the human genome (set of human genes). Researchers study the association between genes and health conditions or personal characteristics like vision, obesity, or behavioral traits. In this part of the study we will be collecting information about your individual genes. We will use this information for our study objectives. In addition, if you agree, the data will be entered into external scientific databases so that it can be broadly shared with other researchers performing other genomic studies. For example, the National Institutes of Health (NIH, an agency of the US federal government) maintains a database called "dbGaP." Databases like this serve as a repository of all kinds of genomic data from studies funded by the NIH and conducted in the US and around the world. The aim of collecting this information in a repository is to allow qualified researchers to look for genetic connections for a range of topics in the future. The information may be used to learn if certain genes are associated with certain traits, diseases and /or treatment effects. Making data broadly available in this way means that your contribution and the data generated in this study could be helpful in advancing other areas of scientific research.

Traditionally used identifying information about you (such as name, phone number, address) will NOT be included in these databases or shared with others. De-identified genomic data generated in this study may be deposited in databases that will be publicly accessible via the Internet. Researches with an approved study may access and utilize your de-identified genetic, genomic and/or health information deposited in the database (dbGAP) after approval by the regulatory authority (NIH). Strict safety measures are in place to protect the privacy of your information. However, because your genetic information is unique to you, there is a small chance that someone could trace it back to you or your family. The risk of this happening is very small, but may grow in the future. Researchers will always have a duty to protect your privacy and keep your information confidential.

You may withdraw consent for research use of genomic data or health information at any time. In this event, data will be withdrawn from any repository, if possible, but data already distributed for research use will not be retrieved.

If you decide not to participate in this part of the study it will not affect your involvement in the main part of the study. This form is designed to allow you to state your preference for this extra participation.

PLEASE TURN OVER

Study number: W \_\_\_\_/\_\_\_

| Please initial boxes if you agree with each statement. |
|--------------------------------------------------------|
|--------------------------------------------------------|

Agree / Consent? Yes No

| 1. | Blood (and if taken, sputum or buccal (chee will be extracted for DNA or RNA which will further our understanding of how asthma detreatment or disease severity. We plan to come and RNA to help identify new genes that man hypotheses of how genes influence treatmen. The information collected in these study significance and there are no plans to common to participants. If you would prefer not to take this study, this will in no way bar you from know whether you would like to take part in the box below. | | |
|---|---|---|---|
| | I agree to take part i | n the genetic analysis | oart of this study |
| 2. | . If you do not wish your data to be shared as described above, you may still take part in this study and your data will not be submitted to an external database. Please indicate below by initialing the appropriate box below whether you consent to the sharing of your data in this way. | | |
| | I consent to my genetic, genomic and/or health information being submitted to an external database and broadly shared with other researchers | | |
| | , | | |
| 3. | <ol> <li>If there are any unused samples remaining after completion of the study, these may<br/>be saved for future asthma related research. Please initial the box below if you are<br/>happy with this.</li> </ol> | | |
| | I agree to have any unused sample(s) to be stored and used for future asthma-related research. | | |
| | Name of Patient Date | | Signature |
| | Name of paragraph taking agreet | | Signature |
| | Name of person taking consent Date | | Signature |

One copy for patient, one for researcher, one to be kept with hospital notes.